CLINICAL TRIAL: NCT05228262
Title: Study on Vascular Function, Sarcopenia and Pain in Treated Postmenopausal Osteoporosis
Brief Title: Vascular Function, Sarcopenia and Pain in Postmenopausal Osteoporosis
Acronym: VASCO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: RBHP 2021 ME_PICKERING; 2021-A02276-35 (Other: ANSM)
Record Dates: First submitted 2022-01-13; First posted 2022-02-08 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2022-01

CONDITIONS: Osteoporosis, Postmenopausal
Keywords: Osteoporosis; Sarcopenia; Cardiovascular; FMD
MeSH Terms: conditions — Osteoporosis, Postmenopausal; Osteoporosis; Sarcopenia

STUDY DESIGN:
Intervention Model Description: Population of postmenopausal women ≥50 years of age with osteoporosis requiring the initiation of antiosteoporotic therapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cohort follow-up (Other): Exploratory study involving functional explorations in longitudinal follow-up, initiated in parallel with a treatment indicated in the patient's usual care and management.
  Interventions: Other: Cohort follow-up

INTERVENTIONS:
Other: Cohort follow-up — * Inclusion medical consultation,
  * Inclusion clinical examination,
  * Collection of biological samples (bone biomarkers, epigenetic biomarkers (microRNA)) and analysis of microbiota and genotyping,
  * Calculation of the Kauppila score on profile spine radiographs by the rheumatologist,
  * Cardiovascular investigations (FMD, "Flow-Mediated Dilation"); measurement of digital volume increase (RHI, "Reactive hyperhemia index"); measurement of microcirculatory perfusion of the skin at the hand (FLD, "Flow Laser Doppler") ; measurement of the stiffness of the main arteries (aorta) by the Pulse Wave Velocity (PWV),
  * Exploration of sarcopenia: questionnaires and tests: SARC-F, SPPB, muscle strength,
  * Quality of life component questionnaires Pittsburgh Sleep (PSQI), Numerical Scale (NS), Brief Pain Inventory (BPI), Hospital Anxiety and Depression scale (HADs), and 36-Item Short Form Survey (SF-36) Quality of Life Questionnaire.

SUMMARY:
This study aims to follow a cohort of osteoporotic patients treated with anti-osteoporotic drugs and to evaluate the impact of these treatments on the osteoporosis-cardiovascular-sarcopenia triad and on pain.

DETAILED DESCRIPTION:
Exploratory study involving functional explorations in longitudinal follow-up, initiated in parallel with a treatment indicated in the patient's usual care and management.

The main objective is the evaluation of the evolution of the vascular and endothelial function.

The secondary objectives are:

1. To study the evolution of cardiovascular parameters,
2. To study the evolution of sarcopenia,
3. To study the evolution of quality of life and pain,
4. To study the evolution of bone remodeling (by creating a collection of biological samples),
5. To study the genetic predisposition of osteoporosis including the confirmation of known genetic markers and the potential identification of new genetic variants involved (by creating a biobank),
6. To study epigenetic biomarkers in the osteoporosis patient population (by creating a biobank),
7. To study the role of the microbiota in osteoporosis patients (by creating a biobank),
8. To study the determinants of the evolution of the studied parameters and to identify trajectories (therapeutic response profiles).

As part of their usual care and management, patients will be diagnosed with osteoporosis and prescribed anti-osteoporotic drugs.

The patients will have six visits: a pre-selection visit that will take place in the Rheumatology Department of the Clermont-Ferrand University Hospital and five visits that will take place in the Clinical Investigation Platform/Clinical Investigation Center (PIC/CIC) Inserm 1405 of the Clermont-Ferrand University Hospital.

Visit 0 - Screening visit and diagnosis of osteoporosis T0-1: Rheumatology Department

During this visit, the investigator physician will perform various examinations and tests usually performed as part of the patient's usual care and management in order to establish a diagnosis of osteoporosis.

These examinations are as follows:

* Bone densitometry less than one year old using Dual energy X-ray Absorptiometry (DXA),
* Bone biological assessment, including the following tests: Complete Blood Count (CBC), platelets, C-Reactive Protein (CRP), urea, creatinine with CKD-EPI clearance calculation, liver enzymes (AST, ALT), serum calcium, serum calcium corrected by albumin, serum phosphorus, serum protein electrophoresis, Thyroid Stimulating Hormone (TSH), 25 OH vitamin D, serum CTX (C-terminal telopeptides of type 1 collagen).

Some patients who require profile radiographs of the spine will have this examination added for the consultation, especially for the evaluation of vertebral fractures if the context justifies it. Other patients will also have these x-rays for the calculation of the abdominal aortic calcification score (Kauppila score) by the rheumatologist.

Body composition will be requested during the bone densitometry evaluation on the DXA machine.

Once the diagnosis of osteoporosis is confirmed, the physician will propose to the eligible patients to participate in this research protocol by explaining the objectives and the course of the study, and give them an information note in order to give them a necessary time of reflection of a maximum of one month, depending on the scheduling of the inclusion visit.

If patients are interested,the investigator physician will prescribe osteoporotic treatment to be started after the V1 (T0) inclusion visit.

Visit 1 - Inclusion visit - T0: PIC/CIC (2 hours)

During this visit, the physician will explain again the objectives and progress of the study with the different tests and questionnaires planned so that the patients can give their informed consent to participate.

During this visit, the following will be performed:

* A medical examination,
* A blood sample in order to obtain a collection of biological samples for the purpose of:

  1. Assess bone biomarkers (osteocalcin, sclerostin, periostin, irisin, N-terminal propeptide of procollagen type 1 (P1NP), Dickkopf-related protein 1 (DKK1) and C-terminal telopeptides of collagen type 1 (CTX)),
  2. Characterize genetic predispositions to osteoporosis,
  3. Characterize epigenetic biomarkers in the osteoporosis patient population by microRNA analysis,
* Stool sampling to obtain a biobank for subsequent microbiota analysis,
* Cardiovascular exploration based on the measurement of the increase in the diameter of the brachial artery (FMD, "Flow-Mediated Dilation"); measurement of the increase in digital volume (RHI, "Reactive Hyperhemia Index") and measurement of the microcirculatory perfusion of the skin at the level of the hand (FLD, "Flow Laser Doppler"), and measurement of the stiffness of the main arteries (aorta) by the technique of Pulse Wave Velocity (PWV) measurement,
* Exploration of sarcopenia: the following questionnaires and tests will be performed: SARC-F (Strength, Assistance with walking, Rising from a chair, Climbing stairs, and Falls) and SPPB (Short Physical Performance Battery),
* Quality of life component questionnaires: Pittsburgh Sleep Quality Index (PSQI), 36-Item Short Form Survey (SF-36), Numerical Pain Scale (NPS), Bref Pain Inventory (BPI), and Hospital Anxiety and Depression scale (HADs).

Visit 2 (T0+1 year) and Visit 4 (T0+3 years): PIC/CIC (1h15)

During this visit, the following examinations, tests and questionnaires will be performed:

* A physical examination,
* A blood and stool sample to obtain a collection of biological samples (bone biomarkers, microRNA and microbiota analyses),
* A cardiovascular exploration with FMD, RHI, FLD and PWV measurements,
* Exploration of sarcopenia: questionnaires and tests SARC-F, SPPB and measurement of muscle function will be performed,
* Quality of life component questionnaires: Pittsburgh Sleep Quality Index (PSQI), SF-36 quality of life questionnaire, Numerical Pain Scale (NPS), Bref Pain Inventory (BPI), and Hospital Anxiety and Depression scale (HADs).

Visit 3 (T0+2 years) and visit 5 (T0+4 years): PIC/CIC (1h30)

During this visit, the following examinations, tests and questionnaires will be performed:

* A physical examination,
* A blood and stool sample to obtain a collection of biological samples (bone biomarkers, microRNA and microbiota analyses),
* A cardiovascular exploration with FMD, RHI, FLD and PWV measurements,
* Exploration of sarcopenia: questionnaires and tests SARC-F, SPPB, measurement of muscle function and DXA with body composition measurement will be performed,
* Quality of life component questionnaires: Pittsburgh Sleep Quality Index (PSQI), SF-36 quality of life questionnaire, Numerical Pain Scale (NPS), Bref Pain Inventory (BPI), and Hospital Anxiety and Depression scale (HADs).

Visit 5 will be the last visit of the study.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 50 years or older with postmenopausal osteoporosis, whether fractured or not, requiring initiation of treatment with antiosteoporotic drugs (bisphosphonates, raloxifene, teriparatide, denosumab and others to come for this indication, including romosozumab), either orally or by injection, as part of their care and management.
* Able to give informed consent to participate in research.
* Affiliation to a Social Security system.

Exclusion Criteria:

* Patient with chronic renal failure, defined as glomerular filtration rate < 30 mL.min-1 estimated by CKD-EPI.
* Patient with a medical and/or surgical history deemed by the investigator or his/her representative to be incompatible with the trial.
* Patient under legal protection or deprived of liberty.
* Refusal to participate.

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-02-15 (Actual); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Endothelial dysfunction measured by FMD (Flow-Mediated Dilation) in patients with anti-osteoporotic treatment | Visit 1: Day 0
  FMD is a non-invasive technique. It was assessed using an ultrasound approach with a high-resolution linear array transducer coupled with computer-assisted analysis software. With this software, changes in the brachial artery could be assessed in real-time through an automated edge detection system. Longitudinal images of the brachial artery were obtained with the transducer fixed on the medial aspect of the dominant arm, approximately 2 cm above the medial epicondyle of the humerus. The transducer was fixed on the arm by a special arm-holding device. The brachial artery diameter was acquired as per a 30 s baseline measure, after which a cuff was placed around forearm (3 cm above wrist) and inflated to 250 mm Hg for 5 min. After cuff deflation, the brachial artery diameter was continuously monitored for 2-4 min to detect the peak artery diameter. FMD was determined as the percentage change in diameter from baseline to peak arterial diameter.
Endothelial dysfunction measured by FMD (Flow-Mediated Dilation) in patients with anti-osteoporotic treatment | Visit 2: Day 0+1 year
  FMD is a non-invasive technique. It was assessed using an ultrasound approach with a high-resolution linear array transducer coupled with computer-assisted analysis software. With this software, changes in the brachial artery could be assessed in real-time through an automated edge detection system. Longitudinal images of the brachial artery were obtained with the transducer fixed on the medial aspect of the dominant arm, approximately 2 cm above the medial epicondyle of the humerus. The transducer was fixed on the arm by a special arm-holding device. The brachial artery diameter was acquired as per a 30 s baseline measure, after which a cuff was placed around forearm (3 cm above wrist) and inflated to 250 mm Hg for 5 min. After cuff deflation, the brachial artery diameter was continuously monitored for 2-4 min to detect the peak artery diameter. FMD was determined as the percentage change in diameter from baseline to peak arterial diameter.
Endothelial dysfunction measured by FMD (Flow-Mediated Dilation) in patients with anti-osteoporotic treatment | Visit 3: Day 0+2 years
  FMD is a non-invasive technique. It was assessed using an ultrasound approach with a high-resolution linear array transducer coupled with computer-assisted analysis software. With this software, changes in the brachial artery could be assessed in real-time through an automated edge detection system. Longitudinal images of the brachial artery were obtained with the transducer fixed on the medial aspect of the dominant arm, approximately 2 cm above the medial epicondyle of the humerus. The transducer was fixed on the arm by a special arm-holding device. The brachial artery diameter was acquired as per a 30 s baseline measure, after which a cuff was placed around forearm (3 cm above wrist) and inflated to 250 mm Hg for 5 min. After cuff deflation, the brachial artery diameter was continuously monitored for 2-4 min to detect the peak artery diameter. FMD was determined as the percentage change in diameter from baseline to peak arterial diameter.
Endothelial dysfunction measured by FMD (Flow-Mediated Dilation) in patients with anti-osteoporotic treatment | Visit 4: Day 0+3 years
  FMD is a non-invasive technique. It was assessed using an ultrasound approach with a high-resolution linear array transducer coupled with computer-assisted analysis software. With this software, changes in the brachial artery could be assessed in real-time through an automated edge detection system. Longitudinal images of the brachial artery were obtained with the transducer fixed on the medial aspect of the dominant arm, approximately 2 cm above the medial epicondyle of the humerus. The transducer was fixed on the arm by a special arm-holding device. The brachial artery diameter was acquired as per a 30 s baseline measure, after which a cuff was placed around forearm (3 cm above wrist) and inflated to 250 mm Hg for 5 min. After cuff deflation, the brachial artery diameter was continuously monitored for 2-4 min to detect the peak artery diameter. FMD was determined as the percentage change in diameter from baseline to peak arterial diameter.
Endothelial dysfunction measured by FMD (Flow-Mediated Dilation) in patients with anti-osteoporotic treatment | Visit 5: Day 0+4 years
  FMD is a non-invasive technique. It was assessed using an ultrasound approach with a high-resolution linear array transducer coupled with computer-assisted analysis software. With this software, changes in the brachial artery could be assessed in real-time through an automated edge detection system. Longitudinal images of the brachial artery were obtained with the transducer fixed on the medial aspect of the dominant arm, approximately 2 cm above the medial epicondyle of the humerus. The transducer was fixed on the arm by a special arm-holding device. The brachial artery diameter was acquired as per a 30 s baseline measure, after which a cuff was placed around forearm (3 cm above wrist) and inflated to 250 mm Hg for 5 min. After cuff deflation, the brachial artery diameter was continuously monitored for 2-4 min to detect the peak artery diameter. FMD was determined as the percentage change in diameter from baseline to peak arterial diameter.

SECONDARY OUTCOMES:
Measurement of digital volume increase by RHI (Reactive hyperhemia index), (Endo-PAT2000; Itamar Medical Ltd, Israel). | Visit 1: Day 0
  RHI is a non-invasive technique. It's measure with a digital plethysmographie device that records pulsatile fluctuations in digital volume at rest and during reactive hyperemia. For the RH-PAT procedure, a peripheral arterial tonometry probe was placed on the right index finger and a control tonometry probe was also placed on the left index finger to eliminate sympathetic nerve effects. In the RH-PAT procedure, the RHI value was calculated as the ratio of the reactive hyperemia between the two hands.
Measurement of digital volume increase by RHI (Reactive hyperhemia index), (Endo-PAT2000; Itamar Medical Ltd, Israel). | Visit 2: Day 0+1 year
  RHI is a non-invasive technique. It's measure with a digital plethysmographie device that records pulsatile fluctuations in digital volume at rest and during reactive hyperemia. For the RH-PAT procedure, a peripheral arterial tonometry probe was placed on the right index finger and a control tonometry probe was also placed on the left index finger to eliminate sympathetic nerve effects. In the RH-PAT procedure, the RHI value was calculated as the ratio of the reactive hyperemia between the two hands.
Measurement of digital volume increase by RHI (Reactive hyperhemia index), (Endo-PAT2000; Itamar Medical Ltd, Israel). | Visit 3: Day 0+2 years
  RHI is a non-invasive technique. It's measure with a digital plethysmographie device that records pulsatile fluctuations in digital volume at rest and during reactive hyperemia. For the RH-PAT procedure, a peripheral arterial tonometry probe was placed on the right index finger and a control tonometry probe was also placed on the left index finger to eliminate sympathetic nerve effects. In the RH-PAT procedure, the RHI value was calculated as the ratio of the reactive hyperemia between the two hands.
Measurement of digital volume increase by RHI (Reactive hyperhemia index), (Endo-PAT2000; Itamar Medical Ltd, Israel). | Visit 4: Day 0+3 years
  RHI is a non-invasive technique. It's measure with a digital plethysmographie device that records pulsatile fluctuations in digital volume at rest and during reactive hyperemia. For the RH-PAT procedure, a peripheral arterial tonometry probe was placed on the right index finger and a control tonometry probe was also placed on the left index finger to eliminate sympathetic nerve effects. In the RH-PAT procedure, the RHI value was calculated as the ratio of the reactive hyperemia between the two hands.
Measurement of digital volume increase by RHI (Reactive hyperhemia index), (Endo-PAT2000; Itamar Medical Ltd, Israel). | Visit 5: Day 0+4 years
  RHI is a non-invasive technique. It's measure with a digital plethysmographie device that records pulsatile fluctuations in digital volume at rest and during reactive hyperemia. For the RH-PAT procedure, a peripheral arterial tonometry probe was placed on the right index finger and a control tonometry probe was also placed on the left index finger to eliminate sympathetic nerve effects. In the RH-PAT procedure, the RHI value was calculated as the ratio of the reactive hyperemia between the two hands.
Microcirculation measurement by FLD (Flow Laser Doppler), PeriFlux® (Perimed) | Visit 1: Day 0
  The Flowmetry by Laser Doppler (FLD) is a non-invasive and validated technique for continuous measurement of the endothelial dependent reactivity in local microcirculation. The flow estimated by this technique is based on the assessment of the Doppler shift of low-power laser light, which is scattered by moving red blood cells. Vascular endothelial function in the micro-vascular compartment is assessed using the laser-doppler system PeriFlux 5010 (Perimed) at the level of the skin of the hands by following the response to a reactive hyperemia induced by a temporary occlusion of the brachial artery (same stimulus as for FMD measurement).
Microcirculation measurement by FLD (Flow Laser Doppler), PeriFlux® (Perimed) | Visit 2: Day 0+1 year
  The Flowmetry by Laser Doppler (FLD) is a non-invasive and validated technique for continuous measurement of the endothelial dependent reactivity in local microcirculation. The flow estimated by this technique is based on the assessment of the Doppler shift of low-power laser light, which is scattered by moving red blood cells. Vascular endothelial function in the micro-vascular compartment is assessed using the laser-doppler system PeriFlux 5010 (Perimed) at the level of the skin of the hands by following the response to a reactive hyperemia induced by a temporary occlusion of the brachial artery (same stimulus as for FMD measurement).
Microcirculation measurement by FLD (Flow Laser Doppler), PeriFlux® (Perimed) | Visit 3: Day 0+2 years
  The Flowmetry by Laser Doppler (FLD) is a non-invasive and validated technique for continuous measurement of the endothelial dependent reactivity in local microcirculation. The flow estimated by this technique is based on the assessment of the Doppler shift of low-power laser light, which is scattered by moving red blood cells. Vascular endothelial function in the micro-vascular compartment is assessed using the laser-doppler system PeriFlux 5010 (Perimed) at the level of the skin of the hands by following the response to a reactive hyperemia induced by a temporary occlusion of the brachial artery (same stimulus as for FMD measurement).
Microcirculation measurement by FLD (Flow Laser Doppler), PeriFlux® (Perimed) | Visit 4: Day 0+3 years
  The Flowmetry by Laser Doppler (FLD) is a non-invasive and validated technique for continuous measurement of the endothelial dependent reactivity in local microcirculation. The flow estimated by this technique is based on the assessment of the Doppler shift of low-power laser light, which is scattered by moving red blood cells. Vascular endothelial function in the micro-vascular compartment is assessed using the laser-doppler system PeriFlux 5010 (Perimed) at the level of the skin of the hands by following the response to a reactive hyperemia induced by a temporary occlusion of the brachial artery (same stimulus as for FMD measurement).
Microcirculation measurement by FLD (Flow Laser Doppler), PeriFlux® (Perimed) | Visit 5: Day 0+4 years
  The Flowmetry by Laser Doppler (FLD) is a non-invasive and validated technique for continuous measurement of the endothelial dependent reactivity in local microcirculation. The flow estimated by this technique is based on the assessment of the Doppler shift of low-power laser light, which is scattered by moving red blood cells. Vascular endothelial function in the micro-vascular compartment is assessed using the laser-doppler system PeriFlux 5010 (Perimed) at the level of the skin of the hands by following the response to a reactive hyperemia induced by a temporary occlusion of the brachial artery (same stimulus as for FMD measurement).
Sphygmocor CPV® (Atcor Medical) large artery stiffness measurement (PWV) | Visit 1: Day 0
  The carotid-femoral Pulse Wave Velocity (PWV) is an established index of arterial stiffness. Pulse, which travels at a higher velocity in stiff arterial vessels, is calculated from measurements of pulse transit time and the distance travelled between the 2 considered recording sites (i.e., carotid artery and femoral artery). The measurements are performed using a validated non-invasive device (SphygmoCor; AtCor Medical Pty. Ltd.) that allows online pulse wave recording and automatic PWV calculation [PWV = distance (m)/transit time (s)].
Sphygmocor CPV® (Atcor Medical) large artery stiffness measurement (PWV) | Visit 2: Day 0+1 year
  The carotid-femoral Pulse Wave Velocity (PWV) is an established index of arterial stiffness. Pulse, which travels at a higher velocity in stiff arterial vessels, is calculated from measurements of pulse transit time and the distance travelled between the 2 considered recording sites (i.e., carotid artery and femoral artery). The measurements are performed using a validated non-invasive device (SphygmoCor; AtCor Medical Pty. Ltd.) that allows online pulse wave recording and automatic PWV calculation [PWV = distance (m)/transit time (s)].
Sphygmocor CPV® (Atcor Medical) large artery stiffness measurement (PWV) | Visit 3: Day 0+2 years
  The carotid-femoral Pulse Wave Velocity (PWV) is an established index of arterial stiffness. Pulse, which travels at a higher velocity in stiff arterial vessels, is calculated from measurements of pulse transit time and the distance travelled between the 2 considered recording sites (i.e., carotid artery and femoral artery). The measurements are performed using a validated non-invasive device (SphygmoCor; AtCor Medical Pty. Ltd.) that allows online pulse wave recording and automatic PWV calculation [PWV = distance (m)/transit time (s)].
Sphygmocor CPV® (Atcor Medical) large artery stiffness measurement (PWV) | Visit 4: Day 0+3 years
  The carotid-femoral Pulse Wave Velocity (PWV) is an established index of arterial stiffness. Pulse, which travels at a higher velocity in stiff arterial vessels, is calculated from measurements of pulse transit time and the distance travelled between the 2 considered recording sites (i.e., carotid artery and femoral artery). The measurements are performed using a validated non-invasive device (SphygmoCor; AtCor Medical Pty. Ltd.) that allows online pulse wave recording and automatic PWV calculation [PWV = distance (m)/transit time (s)].
Sphygmocor CPV® (Atcor Medical) large artery stiffness measurement (PWV) | Visit 5: Day 0+4 years
  The carotid-femoral Pulse Wave Velocity (PWV) is an established index of arterial stiffness. Pulse, which travels at a higher velocity in stiff arterial vessels, is calculated from measurements of pulse transit time and the distance travelled between the 2 considered recording sites (i.e., carotid artery and femoral artery). The measurements are performed using a validated non-invasive device (SphygmoCor; AtCor Medical Pty. Ltd.) that allows online pulse wave recording and automatic PWV calculation [PWV = distance (m)/transit time (s)].
Evaluation of the Abdominal Aorta Calcification (AAC) (Kauppila score) | Preselection visit V0: Day 0-1 month (D0-1)
  The Kauppila score is used to estimate the existence and severity of AAC. This semi-quantitative score is used to assign a score from 0 to 3, depending on the severity of vascular calcification, for the anterior and posterior walls of the aortic vessel wall, opposite each lumbar vertebrae from L1 to L4. A maximum score of 24 is thus obtained.
Evaluation of the Abdominal Aorta Calcification (AAC) (Kauppila score) | Visit 5: Day 0+4 years
  The Kauppila score is used to estimate the existence and severity of AAC. This semi-quantitative score is used to assign a score from 0 to 3, depending on the severity of vascular calcification, for the anterior and posterior walls of the aortic vessel wall, opposite each lumbar vertebrae from L1 to L4. A maximum score of 24 is thus obtained.
Strength, Assistance with walking, Rising from a chair, Climbing stairs, and Falls (SARC-F) questionnaire | Visit 1: Day 0
  Consists of 5 questions and a score higher than 4 suggests the presence of sarcopenia (or age-related muscular dystrophy). On the other hand, if the score is less than or equal to 3, the patient is diagnosed as "non-sarcopenic" but tests must be repeated regularly in clinical practice.
Strength, Assistance with walking, Rising from a chair, Climbing stairs, and Falls (SARC-F) questionnaire | Visit 2: Day 0+1 year
  Consists of 5 questions and a score higher than 4 suggests the presence of sarcopenia (or age-related muscular dystrophy). On the other hand, if the score is less than or equal to 3, the patient is diagnosed as "non-sarcopenic" but tests must be repeated regularly in clinical practice.
Strength, Assistance with walking, Rising from a chair, Climbing stairs, and Falls (SARC-F) questionnaire | Visit 3: Day 0+2 years
  Consists of 5 questions and a score higher than 4 suggests the presence of sarcopenia (or age-related muscular dystrophy). On the other hand, if the score is less than or equal to 3, the patient is diagnosed as "non-sarcopenic" but tests must be repeated regularly in clinical practice.
Strength, Assistance with walking, Rising from a chair, Climbing stairs, and Falls (SARC-F) questionnaire | Visit 4: Day 0+3 years
  Consists of 5 questions and a score higher than 4 suggests the presence of sarcopenia (or age-related muscular dystrophy). On the other hand, if the score is less than or equal to 3, the patient is diagnosed as "non-sarcopenic" but tests must be repeated regularly in clinical practice.
Strength, Assistance with walking, Rising from a chair, Climbing stairs, and Falls (SARC-F) questionnaire | Visit 5: Day 0+4 years
  Consists of 5 questions and a score higher than 4 suggests the presence of sarcopenia (or age-related muscular dystrophy). On the other hand, if the score is less than or equal to 3, the patient is diagnosed as "non-sarcopenic" but tests must be repeated regularly in clinical practice.
Short Physical Performance Battery (SPPB) Questionnaire | Visit 1: Day 0
  The Short Physical Performance Battery is the sum of the scores on three criteria: the balance test, the walking speed test and the chair lift test. This test is used to evaluate the physical performance of an individual. Adding the scores of all the tests gives an overall performance score. A score below 8 is an indicator of risk of sarcopenia (0-6 low performance 7-9, intermediate; 10-12 high).
SPPB Questionnaire | Visit 2: Day 0+1 year
  The Short Physical Performance Battery is the sum of the scores on three criteria: the balance test, the walking speed test and the chair lift test. This test is used to evaluate the physical performance of an individual. Adding the scores of all the tests gives an overall performance score. A score below 8 is an indicator of risk of sarcopenia (0-6 low performance 7-9, intermediate; 10-12 high).
SPPB Questionnaire | Visit 3: Day 0+2 years
  The Short Physical Performance Battery is the sum of the scores on three criteria: the balance test, the walking speed test and the chair lift test. This test is used to evaluate the physical performance of an individual. Adding the scores of all the tests gives an overall performance score. A score below 8 is an indicator of risk of sarcopenia (0-6 low performance 7-9, intermediate; 10-12 high).
SPPB Questionnaire | Visit 4: Day 0+3 years
  The Short Physical Performance Battery is the sum of the scores on three criteria: the balance test, the walking speed test and the chair lift test. This test is used to evaluate the physical performance of an individual. Adding the scores of all the tests gives an overall performance score. A score below 8 is an indicator of risk of sarcopenia (0-6 low performance 7-9, intermediate; 10-12 high).
SPPB Questionnaire | Visit 5: Day 0+4 years
  The Short Physical Performance Battery is the sum of the scores on three criteria: the balance test, the walking speed test and the chair lift test. This test is used to evaluate the physical performance of an individual. Adding the scores of all the tests gives an overall performance score. A score below 8 is an indicator of risk of sarcopenia (0-6 low performance 7-9, intermediate; 10-12 high).
Evaluation of the muscular strength | Visit 1: Day 0
  A dynamometer measures grip strength, which decreases with age and is associated with more sarcopenia and cardiovascular comorbidities. The dynamometer is held in the dominant hand, in a sitting position, elbow bent at 90°, shoulders relaxed and forearm in a neutral position. The measurement is taken twice and the highest value is retained. Muscle strength is low when the grip strength is less than 27kg for men or 16kg for women.
Evaluation of the muscular strength | Visit 2: Day 0+1 year
  A dynamometer measures grip strength, which decreases with age and is associated with more sarcopenia and cardiovascular comorbidities. The dynamometer is held in the dominant hand, in a sitting position, elbow bent at 90°, shoulders relaxed and forearm in a neutral position. The measurement is taken twice and the highest value is retained. Muscle strength is low when the grip strength is less than 27kg for men or 16kg for women.
Evaluation of the muscular strength | Visit 3: Day 0+2 years
  A dynamometer measures grip strength, which decreases with age and is associated with more sarcopenia and cardiovascular comorbidities. The dynamometer is held in the dominant hand, in a sitting position, elbow bent at 90°, shoulders relaxed and forearm in a neutral position. The measurement is taken twice and the highest value is retained. Muscle strength is low when the grip strength is less than 27kg for men or 16kg for women.
Evaluation of the muscular strength | Visit 4: Day 0+3 years
  A dynamometer measures grip strength, which decreases with age and is associated with more sarcopenia and cardiovascular comorbidities. The dynamometer is held in the dominant hand, in a sitting position, elbow bent at 90°, shoulders relaxed and forearm in a neutral position. The measurement is taken twice and the highest value is retained. Muscle strength is low when the grip strength is less than 27kg for men or 16kg for women.
Evaluation of the muscular strength | Visit 5: Day 0+4 years
  A dynamometer measures grip strength, which decreases with age and is associated with more sarcopenia and cardiovascular comorbidities. The dynamometer is held in the dominant hand, in a sitting position, elbow bent at 90°, shoulders relaxed and forearm in a neutral position. The measurement is taken twice and the highest value is retained. Muscle strength is low when the grip strength is less than 27kg for men or 16kg for women.
Body composition measurement on Dual energy X-ray Absorptiometry (DXA) | Preselection visit V0: Day 0-1 month (D0-1)
  Body composition analysis by DXA, and quantification of appendicular muscle mass, is the reference method for the diagnosis of sarcopenia. It consists of measuring the appendicular skeletal mass (ASM), i.e. the muscle mass of the upper and lower limbs, or the ASM index (ASMI = ASM/height2). Sarcopenia is confirmed when the MSA is less than 20kg in men and 15kg in women or when the ASMI is less than 7kg/m2 in men and 5.5kg/m2 in women.
Body composition measurement on Dual energy X-ray Absorptiometry (DXA) | Visit 3: Day 0+2 years
  Body composition analysis by DXA, and quantification of appendicular muscle mass, is the reference method for the diagnosis of sarcopenia. It consists of measuring the appendicular skeletal mass (ASM), i.e. the muscle mass of the upper and lower limbs, or the ASM index (ASMI = ASM/height2). Sarcopenia is confirmed when the MSA is less than 20kg in men and 15kg in women or when the ASMI is less than 7kg/m2 in men and 5.5kg/m2 in women.
Body composition measurement on Dual energy X-ray Absorptiometry (DXA) | Visit 5: Day 0+4 years
  Body composition analysis by DXA, and quantification of appendicular muscle mass, is the reference method for the diagnosis of sarcopenia. It consists of measuring the appendicular skeletal mass (ASM), i.e. the muscle mass of the upper and lower limbs, or the ASM index (ASMI = ASM/height2). Sarcopenia is confirmed when the MSA is less than 20kg in men and 15kg in women or when the ASMI is less than 7kg/m2 in men and 5.5kg/m2 in women.
The Pittsburgh Sleep Quality Index (PSQI) | Visit 1: Day 0
  The PSQI is a self-administered questionnaire with 19 items. It was developed to measure sleep quality in the month prior to the patient interview. This questionnaire includes 7 components: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbance, hypnotic medication use and daytime dysfunction.
  The global score (0 to 21) is obtained by adding the sub-scores of the 7 components, each ranging from 0 to 3 points. In the absence of an answer to one or more questions, the subtotal using this question cannot be calculated and will affect the overall score.
  The higher the overall score, the greater the impairment in sleep quality. An overall score >5 is an indicator of sleep disturbance.
The Pittsburgh Sleep Quality Index (PSQI) | Visit 2: Day 0+1 year
  The PSQI is a self-administered questionnaire with 19 items. It was developed to measure sleep quality in the month prior to the patient interview. This questionnaire includes 7 components: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbance, hypnotic medication use and daytime dysfunction.
  The global score (0 to 21) is obtained by adding the sub-scores of the 7 components, each ranging from 0 to 3 points. In the absence of an answer to one or more questions, the subtotal using this question cannot be calculated and will affect the overall score.
  The higher the overall score, the greater the impairment in sleep quality. An overall score >5 is an indicator of sleep disturbance.
The Pittsburgh Sleep Quality Index (PSQI) | Visit 3: Day 0+2 years
  The PSQI is a self-administered questionnaire with 19 items. It was developed to measure sleep quality in the month prior to the patient interview. This questionnaire includes 7 components: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbance, hypnotic medication use and daytime dysfunction.
  The global score (0 to 21) is obtained by adding the sub-scores of the 7 components, each ranging from 0 to 3 points. In the absence of an answer to one or more questions, the subtotal using this question cannot be calculated and will affect the overall score.
  The higher the overall score, the greater the impairment in sleep quality. An overall score >5 is an indicator of sleep disturbance.
The Pittsburgh Sleep Quality Index (PSQI) | Visit 4: Day 0+3 years
  The PSQI is a self-administered questionnaire with 19 items. It was developed to measure sleep quality in the month prior to the patient interview. This questionnaire includes 7 components: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbance, hypnotic medication use and daytime dysfunction.
  The global score (0 to 21) is obtained by adding the sub-scores of the 7 components, each ranging from 0 to 3 points. In the absence of an answer to one or more questions, the subtotal using this question cannot be calculated and will affect the overall score.
  The higher the overall score, the greater the impairment in sleep quality. An overall score >5 is an indicator of sleep disturbance.
The Pittsburgh Sleep Quality Index (PSQI) | Visit 5: Day 0+4 years
  The PSQI is a self-administered questionnaire with 19 items. It was developed to measure sleep quality in the month prior to the patient interview. This questionnaire includes 7 components: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbance, hypnotic medication use and daytime dysfunction.
  The global score (0 to 21) is obtained by adding the sub-scores of the 7 components, each ranging from 0 to 3 points. In the absence of an answer to one or more questions, the subtotal using this question cannot be calculated and will affect the overall score.
  The higher the overall score, the greater the impairment in sleep quality. An overall score >5 is an indicator of sleep disturbance.
The Brief Pain Inventory Questionnaire (BPI) | Visit 1: Day 0
  This self-assessment scale allows the patient to characterize the pain in terms of its intensity and its psychosocial repercussions by means of 11 scales rated from 0 (no pain or does not bother) to 10 (the most horrible pain you can imagine or completely bothers you).
  The QCD also asks the patient to black out the painful areas on a diagram (front and back) and to put an "S" if the pain is on the surface or a "P" if it is deep. The questionnaire also asks the patient to indicate what treatment or medication he or she is taking for the pain and what percentage improvement has been obtained.
The Brief Pain Inventory Questionnaire (BPI) | Visit 2: Day 0+1 year
  This self-assessment scale allows the patient to characterize the pain in terms of its intensity and its psychosocial repercussions by means of 11 scales rated from 0 (no pain or does not bother) to 10 (the most horrible pain you can imagine or completely bothers you).
  The QCD also asks the patient to black out the painful areas on a diagram (front and back) and to put an "S" if the pain is on the surface or a "P" if it is deep. The questionnaire also asks the patient to indicate what treatment or medication he or she is taking for the pain and what percentage improvement has been obtained.
The Brief Pain Inventory Questionnaire (BPI) | Visit 3: Day 0+2 years
  This self-assessment scale allows the patient to characterize the pain in terms of its intensity and its psychosocial repercussions by means of 11 scales rated from 0 (no pain or does not bother) to 10 (the most horrible pain you can imagine or completely bothers you).
  The QCD also asks the patient to black out the painful areas on a diagram (front and back) and to put an "S" if the pain is on the surface or a "P" if it is deep. The questionnaire also asks the patient to indicate what treatment or medication he or she is taking for the pain and what percentage improvement has been obtained.
The Brief Pain Inventory Questionnaire (BPI) | Visit 4: Day 0+3 years
  This self-assessment scale allows the patient to characterize the pain in terms of its intensity and its psychosocial repercussions by means of 11 scales rated from 0 (no pain or does not bother) to 10 (the most horrible pain you can imagine or completely bothers you).
  The QCD also asks the patient to black out the painful areas on a diagram (front and back) and to put an "S" if the pain is on the surface or a "P" if it is deep. The questionnaire also asks the patient to indicate what treatment or medication he or she is taking for the pain and what percentage improvement has been obtained.
The Brief Pain Inventory Questionnaire (BPI) | Visit 5: Day 0+4 years
  This self-assessment scale allows the patient to characterize the pain in terms of its intensity and its psychosocial repercussions by means of 11 scales rated from 0 (no pain or does not bother) to 10 (the most horrible pain you can imagine or completely bothers you).
  The QCD also asks the patient to black out the painful areas on a diagram (front and back) and to put an "S" if the pain is on the surface or a "P" if it is deep. The questionnaire also asks the patient to indicate what treatment or medication he or she is taking for the pain and what percentage improvement has been obtained.
The numerical pain scale | Visit 1: Day 0
  This scale allows the patient to rate the pain on a scale with a minimum score of 0 (no pain) and a maximum score of 10 (worst pain).
The numerical pain scale | Visit 2: Day 0+1 year
  This scale allows the patient to rate the pain on a scale with a minimum score of 0 (no pain) and a maximum score of 10 (worst pain).
The numerical pain scale | Visit 3: Day 0+2 years
  This scale allows the patient to rate the pain on a scale with a minimum score of 0 (no pain) and a maximum score of 10 (worst pain).
The numerical pain scale | Visit 4: Day 0+3 years
  This scale allows the patient to rate the pain on a scale with a minimum score of 0 (no pain) and a maximum score of 10 (worst pain).
The numerical pain scale | Visit 5: Day 0+4 years
  This scale allows the patient to rate the pain on a scale with a minimum score of 0 (no pain) and a maximum score of 10 (worst pain).
The Hospital Anxiety and Depression Scale (HAD) | Visit 1: Day 0
  It is a self-administered questionnaire completed by the patient and based on the Hamilton scale. The HAD scale is a tool for screening for anxiety and depressive disorders. It includes 14 items rated from 0 to 3. Seven questions relate to anxiety (total A) and seven others to the depressive dimension (total D), thus making it possible to obtain two scores (maximum score for each score = 21).
  To screen for anxiety and depressive symptomatology, the following interpretation can be proposed for each of the scores (A and D): ≤ 7: normal case; 8 to 10: borderline case; ≥ 11: abnormal case.
The Hospital Anxiety and Depression Scale (HAD) | Visit 2: Day 0+1 year
  It is a self-administered questionnaire completed by the patient and based on the Hamilton scale. The HAD scale is a tool for screening for anxiety and depressive disorders. It includes 14 items rated from 0 to 3. Seven questions relate to anxiety (total A) and seven others to the depressive dimension (total D), thus making it possible to obtain two scores (maximum score for each score = 21).
  To screen for anxiety and depressive symptomatology, the following interpretation can be proposed for each of the scores (A and D): ≤ 7: normal case; 8 to 10: borderline case; ≥ 11: abnormal case.
The Hospital Anxiety and Depression Scale (HAD) | Visit 3: Day 0+2 years
  It is a self-administered questionnaire completed by the patient and based on the Hamilton scale. The HAD scale is a tool for screening for anxiety and depressive disorders. It includes 14 items rated from 0 to 3. Seven questions relate to anxiety (total A) and seven others to the depressive dimension (total D), thus making it possible to obtain two scores (maximum score for each score = 21).
  To screen for anxiety and depressive symptomatology, the following interpretation can be proposed for each of the scores (A and D): ≤ 7: normal case; 8 to 10: borderline case; ≥ 11: abnormal case.
The Hospital Anxiety and Depression Scale (HAD) | Visit 4: Day 0+3 years
  It is a self-administered questionnaire completed by the patient and based on the Hamilton scale. The HAD scale is a tool for screening for anxiety and depressive disorders. It includes 14 items rated from 0 to 3. Seven questions relate to anxiety (total A) and seven others to the depressive dimension (total D), thus making it possible to obtain two scores (maximum score for each score = 21).
  To screen for anxiety and depressive symptomatology, the following interpretation can be proposed for each of the scores (A and D): ≤ 7: normal case; 8 to 10: borderline case; ≥ 11: abnormal case.
The Hospital Anxiety and Depression Scale (HAD) | Visit 5: Day 0+4 years
  It is a self-administered questionnaire completed by the patient and based on the Hamilton scale. The HAD scale is a tool for screening for anxiety and depressive disorders. It includes 14 items rated from 0 to 3. Seven questions relate to anxiety (total A) and seven others to the depressive dimension (total D), thus making it possible to obtain two scores (maximum score for each score = 21).
  To screen for anxiety and depressive symptomatology, the following interpretation can be proposed for each of the scores (A and D): ≤ 7: normal case; 8 to 10: borderline case; ≥ 11: abnormal case.
The 36-Item Short Form Survey (SF-36) | Visit 1: Day 0
  The quality of life of patients is assessed by the general questionnaire 36-Item Short Form Survey (SF-36) which can be administered by self or hetero-questionnaire. The SF-36 questionnaire was developed from the Medical Outcome Study, a 149-item questionnaire that was developed to assess how the American healthcare system affects the outcome of care. The SF-36 questionnaire is composed of 36 items and makes it possible to assess the physical and mental health of an individual using eleven questions relating to eight aspects of health: Physical activity, limitations due to physical state, physical pain, perceived health, vitality, life and relationship with others, limitations due to the mental state and mental health. Scores between 0 and 100 are determined. Scores tending towards 100 indicate a better quality of life.
The 36-Item Short Form Survey (SF-36) | Visit 2: Day 0+1 year
  The quality of life of patients is assessed by the general questionnaire 36-Item Short Form Survey (SF-36) which can be administered by self or hetero-questionnaire. The SF-36 questionnaire was developed from the Medical Outcome Study, a 149-item questionnaire that was developed to assess how the American healthcare system affects the outcome of care. The SF-36 questionnaire is composed of 36 items and makes it possible to assess the physical and mental health of an individual using eleven questions relating to eight aspects of health: Physical activity, limitations due to physical state, physical pain, perceived health, vitality, life and relationship with others, limitations due to the mental state and mental health. Scores between 0 and 100 are determined. Scores tending towards 100 indicate a better quality of life.
The 36-Item Short Form Survey (SF-36) | Visit 3: Day 0+2 years
  The quality of life of patients is assessed by the general questionnaire 36-Item Short Form Survey (SF-36) which can be administered by self or hetero-questionnaire. The SF-36 questionnaire was developed from the Medical Outcome Study, a 149-item questionnaire that was developed to assess how the American healthcare system affects the outcome of care. The SF-36 questionnaire is composed of 36 items and makes it possible to assess the physical and mental health of an individual using eleven questions relating to eight aspects of health: Physical activity, limitations due to physical state, physical pain, perceived health, vitality, life and relationship with others, limitations due to the mental state and mental health. Scores between 0 and 100 are determined. Scores tending towards 100 indicate a better quality of life.
The 36-Item Short Form Survey (SF-36) | Visit 4: Day 0+3 years
  The quality of life of patients is assessed by the general questionnaire 36-Item Short Form Survey (SF-36) which can be administered by self or hetero-questionnaire. The SF-36 questionnaire was developed from the Medical Outcome Study, a 149-item questionnaire that was developed to assess how the American healthcare system affects the outcome of care. The SF-36 questionnaire is composed of 36 items and makes it possible to assess the physical and mental health of an individual using eleven questions relating to eight aspects of health: Physical activity, limitations due to physical state, physical pain, perceived health, vitality, life and relationship with others, limitations due to the mental state and mental health. Scores between 0 and 100 are determined. Scores tending towards 100 indicate a better quality of life.
The 36-Item Short Form Survey (SF-36) | Visit 5: Day 0+4 years
  The quality of life of patients is assessed by the general questionnaire 36-Item Short Form Survey (SF-36) which can be administered by self or hetero-questionnaire. The SF-36 questionnaire was developed from the Medical Outcome Study, a 149-item questionnaire that was developed to assess how the American healthcare system affects the outcome of care. The SF-36 questionnaire is composed of 36 items and makes it possible to assess the physical and mental health of an individual using eleven questions relating to eight aspects of health: Physical activity, limitations due to physical state, physical pain, perceived health, vitality, life and relationship with others, limitations due to the mental state and mental health. Scores between 0 and 100 are determined. Scores tending towards 100 indicate a better quality of life.
Sclerostin dosage | Visit 1: Day 0
  The dosage of slerostin (ng/ml) will be performed in order to evaluate bone remodeling. For this purpose, a blood sample will be taken using 5 mL dry tubes
Sclerostin dosage | Visit 2: Day 0+1 year
  The dosage of slerostin (ng/ml) will be performed in order to evaluate bone remodeling. For this purpose, a blood sample will be taken using 5 mL dry tubes
Sclerostin dosage | Visit 3: Day 0+2 years
  The dosage of slerostin (ng/ml) will be performed in order to evaluate bone remodeling. For this purpose, a blood sample will be taken using 5 mL dry tubes
Sclerostin dosage | Visit 4: Day 0+3 years
  The dosage of slerostin (ng/ml) will be performed in order to evaluate bone remodeling. For this purpose, a blood sample will be taken using 5 mL dry tubes
Sclerostin dosage | Visit 5: Day 0+4 years
  The dosage of slerostin (ng/ml) will be performed in order to evaluate bone remodeling. For this purpose, a blood sample will be taken using 5 mL dry tubes
Osteocalcin dosage | Visit 1: Day 0
  The dosage of osteocalcin (ng/ml) will be performed in order to evaluate bone remodeling. For this purpose, a blood sample will be taken using 5 mL dry tubes
Osteocalcin dosage | Visit 2: Day 0+1 year
  The dosage of osteocalcin (ng/ml) will be performed in order to evaluate bone remodeling. For this purpose, a blood sample will be taken using 5 mL dry tubes
Osteocalcin dosage | Visit 3: Day 0+2 years
  The dosage of osteocalcin (ng/ml) will be performed in order to evaluate bone remodeling. For this purpose, a blood sample will be taken using 5 mL dry tubes
Osteocalcin dosage | Visit 4: Day 0+3 years
  The dosage of osteocalcin (ng/ml) will be performed in order to evaluate bone remodeling. For this purpose, a blood sample will be taken using 5 mL dry tubes
Osteocalcin dosage | Visit 5: Day 0+4 years
  The dosage of osteocalcin (ng/ml) will be performed in order to evaluate bone remodeling. For this purpose, a blood sample will be taken using 5 mL dry tubes
Periostin dosage | Visit 1: Day 0
  The dosage of periostin (ng/ml) will be performed in order to evaluate bone remodeling. For this purpose, a blood sample will be taken using 5 mL dry tubes
Periostin dosage | Visit 2: Day 0+1 year
  The dosage of periostin (ng/ml) will be performed in order to evaluate bone remodeling. For this purpose, a blood sample will be taken using 5 mL dry tubes
Periostin dosage | Visit 3: Day 0+2 years
  The dosage of periostin (ng/ml) will be performed in order to evaluate bone remodeling. For this purpose, a blood sample will be taken using 5 mL dry tubes
Periostin dosage | Visit 4: Day 0+3 years
  The dosage of periostin (ng/ml) will be performed in order to evaluate bone remodeling. For this purpose, a blood sample will be taken using 5 mL dry tubes
Periostin dosage | Visit 5: Day 0+4 years
  The dosage of periostin (ng/ml) will be performed in order to evaluate bone remodeling. For this purpose, a blood sample will be taken using 5 mL dry tubes
Irisin dosage | Visit 1: Day 0
  The dosage of irisin (ng/ml) will be performed in order to evaluate bone remodeling. For this purpose, a blood sample will be taken on 4 mL heparin tube for irisin dosage.
Irisin dosage | Visit 2: Day 0+1 year
  The dosage of irisin (ng/ml) will be performed in order to evaluate bone remodeling. For this purpose, a blood sample will be taken on 4 mL heparin tube for irisin dosage.
Irisin dosage | Visit 3: Day 0+2 years
  The dosage of irisin (ng/ml) will be performed in order to evaluate bone remodeling. For this purpose, a blood sample will be taken on 4 mL heparin tube for irisin dosage.
Irisin dosage | Visit 4: Day 0+3 years
  The dosage of irisin (ng/ml) will be performed in order to evaluate bone remodeling. For this purpose, a blood sample will be taken on 4 mL heparin tube for irisin dosage.
Irisin dosage | Visit 5: Day 0+4 years
  The dosage of irisin (ng/ml) will be performed in order to evaluate bone remodeling. For this purpose, a blood sample will be taken on 4 mL heparin tube for irisin dosage.
N-terminal propeptide of procollagen type 1 (P1NP) dosage | Visit 1: Day 0
  The dosage of N-terminal propeptide of procollagen type 1 (P1NP) (µg/l) will be performed in order to evaluate bone remodeling. For this purpose, a blood sample will be taken using 5 mL dry tubes
N-terminal propeptide of procollagen type 1 (P1NP) dosage | Visit 2: Day 0+1 year
  The dosage of N-terminal propeptide of procollagen type 1 (P1NP) (µg/l) will be performed in order to evaluate bone remodeling. For this purpose, a blood sample will be taken using 5 mL dry tubes
N-terminal propeptide of procollagen type 1 (P1NP) dosage | Visit 3: Day 0+2 years
  The dosage of N-terminal propeptide of procollagen type 1 (P1NP) (µg/l) will be performed in order to evaluate bone remodeling. For this purpose, a blood sample will be taken using 5 mL dry tubes
N-terminal propeptide of procollagen type 1 (P1NP) dosage | Visit 4: Day 0+3 years
  The dosage of N-terminal propeptide of procollagen type 1 (P1NP) (µg/l) will be performed in order to evaluate bone remodeling. For this purpose, a blood sample will be taken using 5 mL dry tubes
N-terminal propeptide of procollagen type 1 (P1NP) dosage | Visit 5: Day 0+4 years
  The dosage of N-terminal propeptide of procollagen type 1 (P1NP) (µg/l) will be performed in order to evaluate bone remodeling. For this purpose, a blood sample will be taken using 5 mL dry tubes
Dickkopf-related protein 1 (DKK1) dosage | Visit 1: Day 0
  The dosage of Dickkopf-related protein 1 (DKK1) (ng/ml) will be performed in order to evaluate bone remodeling. For this purpose, a blood sample will be taken using 5 mL dry tubes
Dickkopf-related protein 1 (DKK1) dosage | Visit 2: Day 0+1 year
  The dosage of Dickkopf-related protein 1 (DKK1) (ng/ml) will be performed in order to evaluate bone remodeling. For this purpose, a blood sample will be taken using 5 mL dry tubes
Dickkopf-related protein 1 (DKK1) dosage | Visit 3: Day 0+2 years
  The dosage of Dickkopf-related protein 1 (DKK1) (ng/ml) will be performed in order to evaluate bone remodeling. For this purpose, a blood sample will be taken using 5 mL dry tubes
Dickkopf-related protein 1 (DKK1) dosage | Visit 4: Day 0+3 years
  The dosage of Dickkopf-related protein 1 (DKK1) (ng/ml) will be performed in order to evaluate bone remodeling. For this purpose, a blood sample will be taken using 5 mL dry tubes
Dickkopf-related protein 1 (DKK1) dosage | Visit 5: Day 0+4 years
  The dosage of Dickkopf-related protein 1 (DKK1) (ng/ml) will be performed in order to evaluate bone remodeling. For this purpose, a blood sample will be taken using 5 mL dry tubes
C-terminal telopeptides of collagen type 1 (CTX) dosage | Visit 1: Day 0
  The dosage of C-terminal telopeptides of collagen type 1 (CTX) (ng/ml) will be performed in order to evaluate bone remodeling. For this purpose, a blood sample will be taken using 5 mL dry tubes
C-terminal telopeptides of collagen type 1 (CTX) dosage | Visit 2: Day 0+1 year
  The dosage of C-terminal telopeptides of collagen type 1 (CTX) (ng/ml) will be performed in order to evaluate bone remodeling. For this purpose, a blood sample will be taken using 5 mL dry tubes
C-terminal telopeptides of collagen type 1 (CTX) dosage | Visit 3: Day 0+2 years
  The dosage of C-terminal telopeptides of collagen type 1 (CTX) (ng/ml) will be performed in order to evaluate bone remodeling. For this purpose, a blood sample will be taken using 5 mL dry tubes
C-terminal telopeptides of collagen type 1 (CTX) dosage | Visit 4: Day 0+3 years
  The dosage of C-terminal telopeptides of collagen type 1 (CTX) (ng/ml) will be performed in order to evaluate bone remodeling. For this purpose, a blood sample will be taken using 5 mL dry tubes
C-terminal telopeptides of collagen type 1 (CTX) dosage | Visit 5: Day 0+4 years
  The dosage of C-terminal telopeptides of collagen type 1 (CTX) (ng/ml) will be performed in order to evaluate bone remodeling. For this purpose, a blood sample will be taken using 5 mL dry tubes
Distribution of gene polymorphisms using OpenArray technology | Visit 1: Day 0
  Blood sampling: 4 aliquots of 1 ml will be taken from the whole blood sample on EDTA tube, then frozen at -80°C in the premises of the PIC/CIC Inserm 1405, Clermont-Ferrand, France for subsequent analysis.
MicroRNA analysis using OpenArray technology | Visit 1: Day 0
  Blood sampling: 1 EDTA tube of 6 ml will be collected for microRNA. The tube will then be centrifuged and 6 aliquots of 0.5 ml will be prepared (centrifugation 2500G/ 10 min/4°C) then frozen and stored at - 80°C in the premises of the PIC/CIC Inserm 1405, Clermont-Ferrand, France for subsequent analysis.
MicroRNA analysis using OpenArray technology | Visit 2: Day 0+1 year
  Blood sampling: 1 EDTA tube of 6 ml will be collected for microRNA. The tube will then be centrifuged and 6 aliquots of 0.5 ml will be prepared (centrifugation 2500G/ 10 min/4°C) then frozen and stored at - 80°C in the premises of the PIC/CIC Inserm 1405, Clermont-Ferrand, France for subsequent analysis.
MicroRNA analysis using OpenArray technology | Visit 3: Day 0+2 years
  Blood sampling: 1 EDTA tube of 6 ml will be collected for microRNA. The tube will then be centrifuged and 6 aliquots of 0.5 ml will be prepared (centrifugation 2500G/ 10 min/4°C) then frozen and stored at - 80°C in the premises of the PIC/CIC Inserm 1405, Clermont-Ferrand, France for subsequent analysis.
MicroRNA analysis using OpenArray technology | Visit 4: Day 0+3 years
  Blood sampling: 1 EDTA tube of 6 ml will be collected for microRNA. The tube will then be centrifuged and 6 aliquots of 0.5 ml will be prepared (centrifugation 2500G/ 10 min/4°C) then frozen and stored at - 80°C in the premises of the PIC/CIC Inserm 1405, Clermont-Ferrand, France for subsequent analysis.
MicroRNA analysis using OpenArray technology | Visit 5: Day 0+4 years
  Blood sampling: 1 EDTA tube of 6 ml will be collected for microRNA. The tube will then be centrifuged and 6 aliquots of 0.5 ml will be prepared (centrifugation 2500G/ 10 min/4°C) then frozen and stored at - 80°C in the premises of the PIC/CIC Inserm 1405, Clermont-Ferrand, France for subsequent analysis.
Study of the microbiota | Visit 1: Day 0
  Stool sampling in order to study the microbiota. The patient must collect the stool at each visit by following the technical instructions described in the explanatory leaflet that will be provided. She must then respect the procedure for the conservation and transport of the stool described in this document. The samples will be stored at the PIC/ CIC Inserm 1405, Clermont-Ferrand, Franced for subsequent analysis.
Study of the microbiota | Visit 2: Day 0+1 year
  Stool sampling in order to study the microbiota. The patient must collect the stool at each visit by following the technical instructions described in the explanatory leaflet that will be provided. She must then respect the procedure for the conservation and transport of the stool described in this document. The samples will be stored at the PIC/ CIC Inserm 1405, Clermont-Ferrand, Franced for subsequent analysis.
Study of the microbiota | Visit 3: Day 0+2 years
  Stool sampling in order to study the microbiota. The patient must collect the stool at each visit by following the technical instructions described in the explanatory leaflet that will be provided. She must then respect the procedure for the conservation and transport of the stool described in this document. The samples will be stored at the PIC/ CIC Inserm 1405, Clermont-Ferrand, Franced for subsequent analysis.
Study of the microbiota | Visit 4: Day 0+3 years
  Stool sampling in order to study the microbiota. The patient must collect the stool at each visit by following the technical instructions described in the explanatory leaflet that will be provided. She must then respect the procedure for the conservation and transport of the stool described in this document. The samples will be stored at the PIC/ CIC Inserm 1405, Clermont-Ferrand, Franced for subsequent analysis.
Study of the microbiota | Visit 5: Day 0+4 years
  Stool sampling in order to study the microbiota. The patient must collect the stool at each visit by following the technical instructions described in the explanatory leaflet that will be provided. She must then respect the procedure for the conservation and transport of the stool described in this document. The samples will be stored at the PIC/ CIC Inserm 1405, Clermont-Ferrand, Franced for subsequent analysis.
Identification of predictive factors of treatment effectiveness according to variations in vascular and endothelial function parameters and pain, which will be studied first as quantitative parameters and then as categorical data. | Through study completion, an average of 1 year
  This parameter will be evaluated according to a statiscal method on all the data collected throughout the study. This statistical method will allow to obtain different trajectories corresponding to therapeutic response profile.

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Eva Pickering, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France